CLINICAL TRIAL: NCT00023322
Title: Treatment of Chronic Delta Hepatitis With Pegylated Interferon
Brief Title: Pegylated Interferon to Treat Chronic Hepatitis D
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 010247; 01-DK-0247 (Other: National Institutes of Health)
Record Dates: First submitted 2001-09-03; First posted 2001-09-03 (Estimated); Results first posted 2013-07-10 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2013-07

CONDITIONS: Hepatitis D
Keywords: Cirrhosis; Chronic Hepatitis; Alpha Interferon; Hepatitis D Virus; Delta Hepatitis; Viral Hepatitis; Antiviral Agents; Hepatitis D; HDV; Liver; Hepatitis
MeSH Terms: conditions — Hepatitis D; Fibrosis; Hepatitis, Chronic; Hepatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Peginterferon Alpha-2a (Experimental): Patients with hepatitis D virus (HDV) infection are treated with pegylated alpha interferon therapy for 3 years. The dose of the drug is 180 mcg/week.
  Interventions: Drug: Peginterferon Alpha-2a

INTERVENTIONS:
Drug: Peginterferon Alpha-2a — Treatment

SUMMARY:
This study will evaluate the safety and effectiveness of a long-acting form of alpha interferon called pegylated interferon in treating hepatitis D virus (HDV) infection. HDV only infects people who already have hepatitis B infection. HDV is often severe and progressive. Alpha interferon is the standard treatment for HDV, given by injection once a day or three times a week for up to 12 months. However, this treatment does not work for everyone, and those who respond usually relapse when the drug is stopped. The sustained-release form of the drug, pegylated interferon, is given just once a week. Pegylated interferon is more effective than standard interferon in hepatitis C patients, with patients experiencing longer-term improvement. This study will evaluate the effects of pegylated interferon on hepatitis D and hepatitis B. It will determine whether long-term therapy with this drug improves inflammation and scarring of the liver, thereby delaying or reversing cirrhosis, and whether the improvement can be maintained.

Patients with chronic hepatitis D over 6 years old may be eligible for this study. Participants will have a medical evaluation, including a history and physical examination, blood tests, routine urinalysis and 24-hour urine collection. Chest X-ray, electrocardiogram, abdominal ultrasound and liver biopsy will be done if these tests have not been done within the last year. In addition, depending on their age and individual health status, some patients may have exercise stress testing, an eye examination, hearing test, and psychiatric consultation. All patients will fill out a health-related quality of life questionnaire.

Patients will receive pegylated interferon by injection once a week and have blood tests to measure the effects of treatment on the liver and on HBV and HDV levels. The medical examination and liver biopsy will be repeated at the end of 12 months. Patients who improved with treatment may continue therapy long-term. Medical evaluations and liver biopsies will be repeated at 3 years and at 5 years.

DETAILED DESCRIPTION:
We propose to treat between 10 and 20 patients with chronic delta hepatitis with pegylated alpha interferon for up to five years. Patients with chronic delta hepatitis with raised serum aminotransferases, HBsAg and HDV RNA in serum, and moderate-to-severe chronic hepatitis on liver biopsy with HDV antigen will be enrolled. Patients will be monitored for at least three months with regular testing for ALT levels and will undergo admission for a thorough medical evaluation, portal pressure measurement and percutaneous liver biopsy before treatment. Pegylated interferon will then be started in a dose of 180 mcg weekly. At each clinic visit, patients will be questioned about side effects and symptoms and have blood taken for complete blood counts and routine liver tests (ALT, AST, alkaline phosphatase, direct and total bilirubin, and albumin). At 12-24 week intervals patients will undergo a physical examination and be tested for HBsAg, anti-HBs, HDV RNA, and prothrombin time. The dose of pegylated interferon will be adjusted based upon side effects and changes in ALT levels, aiming for optimal suppression of ALT elevations with acceptable tolerance. At 48 weeks (one year) and every 96 weeks (two years) thereafter, patients will be readmitted to the NIH Clinical Center for repeat thorough medical evaluation, portal pressure measurement and liver biopsy. The primary endpoint of therapy will be improvements in hepatic histology on liver biopsy done after 3 years of pegylated alpha interferon therapy. Several secondary endpoints will be measured, including changes in HDV RNA, loss of HBsAg, HDV staining in the liver biopsy, ALT levels, changes in portal pressures, quality of life, all at 1.3 and 5 years, and hepatic histology at 1 and 5 years. Patients will be maintained on pegylated interferon if it is adequately tolerated and there is an adequate "histological response," as defined by at least 3 point improvement in inflammatory score or 1 point improvement in fibrosis score of the HAI at each liver biopsy. Therapy will be stopped for: (1) intolerance to alpha interferon (which will be carefully defined), (2) lack of improvement in hepatic histology after 1, 3, or 5 years of therapy (histological nonresponse), or (3) a "complete response," i.e. loss of HDV RNA and HBsAg and development of anti-HBs.

ELIGIBILITY:
* INCLUSION CRITERIA:

Age greater than or equal to 18 years, male or female

Serum alanine or aspartate aminotransferase activities that are above the upper limit of normal (ALT greater than 41 or AST greater than 31 U/L) on an average of three determinations taken during the previous 6 months. The mean of the three determinations will be defined as 'baseline' levels.

Presence of anti-HDV in serum.

Evidence of chronic hepatitis on liver biopsy done within the previous 12 months with a necroinflammatory score in histology activity index of at least 5 (out of a maximum of 18) and at least 1 for hepatic fibrosis (out of a maximum of 6).

Presence of HDV antigen in liver tissue.

Written informed consent.

Previous standard alpha interferon or other antiviral activity will not exclude patients.

Active HBV replication will not exclude patients.

All ethnicities.

Patients will need to meet the first six entry criteria to enroll.

EXCLUSION CRITERIA:

Decompensated liver disease, as marked by bilirubin greater than 4 mg%, albumin less than 3.0 gm%, prothrombin time greater than 2 sec prolonged, or history of bleeding esophageal varices, ascites or hepatic encephalopathy. Patients with ALT levels greater than 1000 U/L (greater than 25 times ULN) will not be enrolled but may be followed until three determinations are below this level.

Pregnancy or, in women of child-bearing potential or in spouses of such women, inability to practice adequate contraception defined as vasectomy in men, tubal ligation in women, or use of condoms and spermicide, or birth control pills, or an intrauterine device, or Depo-Provera, or Norplant.

Significant systemic or major illnesses other than liver disease, including, but not limited to, congestive heart failure, renal failure (creatinine clearance less than 50 ml/min), organ transplantation, serious psychiatric disease or depression (only if felt to be at high risk by the NIH psychiatric consultation service), and angina pectoris.

Immunosuppressive therapy within the last 6 months.

Evidence of another form of liver disease in addition to viral hepatitis (for example autoimmune liver disease, Wilson's disease, alcoholic liver disease, hemochromatosis, and alpha-1-antitrypsin deficiency).

Any evidence of coronary artery disease or cerebral vascular disease, including abnormalities on exercise stress testing in patients with defined risk factors who will be screened for evidence of underlying coronary artery disease.

Active substance abuse, such as alcohol, inhaled or injection drugs within the previous year.

Evidence of hepatocellular carcinoma; either alphafetoprotein (AFP) levels greater than 200 ng/ml (normal less than 9 ng/ml) and/or ultrasound (or other imaging study) demonstrating a mass suggestive of liver cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2001-08; Primary Completion 2012-05 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theo Heller, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Verme G, Brunetto MR, Oliveri F, Baldi M, Forzani B, Piantino P, Ponzetto A, Bonino F. Role of hepatitis delta virus infection in hepatocellular carcinoma. Dig Dis Sci. 1991 Aug;36(8):1134-6. doi: 10.1007/BF01297460. PMID 1650690
- [Background] Rizzetto M, Ponzetto A, Forzani I. Hepatitis delta virus as a global health problem. Vaccine. 1990 Mar;8 Suppl:S10-4; discussion S21-3. doi: 10.1016/0264-410x(90)90207-3. PMID 2183511
- [Background] Rizzetto M, Verme G, Recchia S, Bonino F, Farci P, Arico S, Calzia R, Picciotto A, Colombo M, Popper H. Chronic hepatitis in carriers of hepatitis B surface antigen, with intrahepatic expression of the delta antigen. An active and progressive disease unresponsive to immunosuppressive treatment. Ann Intern Med. 1983 Apr;98(4):437-41. doi: 10.7326/0003-4819-98-4-437. PMID 6340574
- [Derived] Hercun J, Kim GE, Da BL, Rotman Y, Kleiner DE, Chang R, Glenn JS, Hoofnagle JH, Koh C, Heller T. Durable virological response and functional cure of chronic hepatitis D after long-term peginterferon therapy. Aliment Pharmacol Ther. 2021 Jul;54(2):176-182. doi: 10.1111/apt.16408. Epub 2021 May 28. PMID 34048594
- [Derived] Kefalakes H, Koh C, Sidney J, Amanakis G, Sette A, Heller T, Rehermann B. Hepatitis D Virus-Specific CD8+ T Cells Have a Memory-Like Phenotype Associated With Viral Immune Escape in Patients With Chronic Hepatitis D Virus Infection. Gastroenterology. 2019 May;156(6):1805-1819.e9. doi: 10.1053/j.gastro.2019.01.035. Epub 2019 Jan 18. PMID 30664876
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2001-DK-0247.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between October 2002 and June 2006, 13 patients were recruited into the study. The location is NIH clinical center.
Period: Overall Study
Arm/Group | Peginterferon Alpha-2a
Started | 13
Completed | 12
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Peginterferon Alpha-2a
Number analyzed (Participants) | 13
Age Continuous [Median (Full Range); unit: years] | 42 [18 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 13
Estimated duration of the disease [Median (Full Range); unit: years] — Estimated duration of the HDV infection
  years | 25 [7 to 35]
ALT [Median (Full Range); unit: IU/L] — alanine aminotransferase
  IU/L | 141 [31 to 506]
Infection source [Number; unit: participants]
  IV Drug Abuse | 6
  Sexual | 2
  Transfusion | 2
  Endemic Region | 5
HDV-RNA [Mean (Standard Deviation); unit: Log10 Genome Equivalent/ml] — hepatitis D virus RNA
  Log10 Genome Equivalent/ml | 6.7 (1.2)
HBsAg [Mean (Standard Deviation); unit: Log10 IU/ml] | 3.7 (0.6)
HBV-DNA [Median (Full Range); unit: Log10 IU/ml] — hepatitis B virus DNA
  Log10 IU/ml | 2.9 [2 to 49]
Fibrosis (Ishak score) [Median (Full Range); unit: Scores on a scale] — Possible range of Ishak score is 0 to 6. Higher values indicate worse outcome.
  Scores on a scale | 3 [3 to 6]

OUTCOME MEASURES:

1. Primary Outcome: Histological Response at 3 Years
Description: Histological response is defined as at least 3 point improvement in inflammatory score or 1 point improvement in fibrosis score of the HAI at each liver biopsy.
Time Frame: 3 years
Population: Intention to treat
Measure: Number; unit: participants
Arm/Group | Peginterferon Alpha-2a
Number analyzed (Participants) | 12
participants | 6

2. Secondary Outcome: Histological Response at 5 Years
Description: as for outcome 1
Time Frame: 5 years
Measure: Number; unit: participants
Arm/Group | Peginterferon Alpha-2a
Number analyzed (Participants) | 12
participants | 6

ADVERSE EVENTS:
Arm/Group | Peginterferon Alpha-2a
Serious Adverse Events (participants affected / at risk) | 1/12
Other Adverse Events (participants affected / at risk) | 3/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peginterferon Alpha-2a (N=12)
Death (Hepatobiliary disorders) | 1 (1) — hepatocellular carcinoma
Death (Hepatobiliary disorders) | 1 (1) — hepatic decompensation secondary to herpes colitis
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peginterferon Alpha-2a (N=12)
soft tissue infection (Skin and subcutaneous tissue disorders) | 1 (1)
autoinflammatory syndrome (Infections and infestations) | 1 (1)
subarachnoid hemorrhage (Blood and lymphatic system disorders) | 1 (1) — subarachnoid hemorrhage from an arteriovenous malformation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes